CLINICAL TRIAL: NCT05540457
Title: Evaluation of Non-Invasive Continuous vs Intermittent BloodPressure Monitors in Maintenance Dialysis
Brief Title: Evaluation of Non-Invasive Continuous vs Intermittent BloodPressure Monitors in Maintenance Dialysis (BP Dialysis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Outset Medical (Industry); CareTaker Medical LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-01
Record Dates: First submitted 2022-08-10; First posted 2022-09-14 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: End Stage Renal Disease; End Stage Renal Disease on Dialysis; Dialysis Hypotension; Dialysis Induced Hypertension
Keywords: Tablo; Outset Medical, Inc.; Caretaker Medical, LLC; VitalStream; ESKD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Non-Invasive Blood Pressure (NIPB)Monitors (Experimental): NIPB Tablo Brachial Cuff (Intermittent): Will be placed contralateral to the access arm. Blood pressure measurements will be collected pre-dialysis, every 30minutes during dialysis, and post-dialysis.
  VitalStream Monitor (Continuous):A cuff will be applied to the middlefinger ipsilateral to the accessarm. Blood pressuremeasurements will be collectedpre-dialysis, continuously duringdialysis, and post-dialysis.
  Interventions: Device: Intermittent Non-InvasiveBlood Pressure Monitor

INTERVENTIONS:
Device: Intermittent Non-InvasiveBlood Pressure Monitor — Brachial cuff integrated with theTablo Hemodialysis System. Cuffwill be placed contralateral to theaccess arm, with measurementscollected pre-dialysis, every 30minutes during dialysis, and post-dialysis.
  Device: Continuous Non-InvasiveBlood Pressure Monitor VitalStream Monitor. Finger cuffwill be placed ipsilateral to theaccess arm, with measurementscollected pre-dialysis,continuously during dialysis, andpost-dialysis.

SUMMARY:
Prospective, single center, open label, non-randomized, post-market study of the Tablo Hemodialysis System and VitalStream Monitor in participants with End-Stage KidneyDisease undergoing In-Center Hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years of age and has provided informed consent and has signed a Health Insurance Portability and Accountability Act of 1996 (HIPAA) compliant authorization statement.
* Participant weighs ≥ 34kg.
* Participant has end stage kidney disease (ESKD) adequately treated by maintenance dialysis.

Exclusion Criteria:

* Participant has lack of perfusion of the digitalarteries and arterioles in the lower arm and hand.
* The Non-Invasive Blood Pressure (NIPB) monitorcuffs (finger and/or brachial) are unable to becorrectly sized to the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Non-invasive Blood Pressure Monitor (NIPB) Measurements | 7 days from start of participation
  Correlation of BP measurements (e.g., systolic, diastolic, mean arterial,and pulse pressures) between NIPB monitors.

SECONDARY OUTCOMES:
Intradialytic Blood Pressure Events | 7 days from start of participation
  Summary of observed intradialytic BP events (hypertensive andhypotensive)
Participant Preference for the Non-invasive Blood Pressure Monitor (NIPB) | 7 days from start of participation
  Participant Preference Questionnaire (PPQ)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Liu, MD, Principal Investigator — The Rogosin Institute, Inc.
Locations (1):
- The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No